CLINICAL TRIAL: NCT03581214
Title: Intrapartum Maternal Oxygen Supplementation: Effects on the Mother and Neonate
Acronym: O2P2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Nandini Raghuraman, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201805045; 1K23HD098315-01A1 (NIH)
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Intrauterine Resuscitation
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Room air (Active Comparator): Room air (no mask)
  Interventions: Other: No oxygen
- Oxygen (Placebo Comparator): 10L/min Oxygen by facemask
  Interventions: Other: Oxygen

INTERVENTIONS:
Other: No oxygen — No facemask, room air only
  Other Names: Room air
  Arms: Room air
Other: Oxygen — 10Liters/minute oxygen by facemask
  Arms: Oxygen

SUMMARY:
Approximately 2/3 of laboring women receive supplemental oxygen (O2) in an attempt to reverse perceived fetal hypoxia on electronic fetal monitoring (EFM). O2 supplementation is most commonly used in patients with Category II EFM, a class of EFM patterns designed in part to identify fetal acidemia. This liberal use of O2 in laboring patients is concerning because hyperoxygenation in infants is associated with adverse outcomes including retinopathy and abnormal neurodevelopment. Furthermore, excess O2 exposure is linked to free radical generation and subsequent oxidative cell damage. This calls for a closer look at the safety of intrauterine O2 exposure. The proposed project explores potential mechanisms for harm with maternal O2 supplementation in laboring patients with Category II EFM. Specifically, this project will determine the effect of O2, compared to room air (RA), on umbilical cord and maternal levels of malondialdehyde (MDA) and 4-hydroxynonenal (4-HNE), markers of free radical-induced oxidative stress. The study will also explore the correlation between urinary and blood markers of oxidative stress. Banked specimens will be used to investigate the potential effect of peripartum O2 exposure on placental oxidative stress in the future.

ELIGIBILITY:
Inclusion Criteria:

* Singleton
* Gestational age ≥37 weeks
* Spontaneous labor or induction of labor
* English speaking
* Ability to give informed consent

Exclusion Criteria:

* Major fetal anomaly
* Multiple gestation
* Category III electronic fetal monitoring
* Maternal hypoxia
* Preeclampsia
* Intrauterine growth restriction
* Pregestational diabetes
* Tobacco use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is in pregnant females only
Enrollment: 910 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2024-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 910 patients were enrolled. Of these, 698 did not get randomized. This was mostly because they did not ultimately meet randomization criteria (N=669), research staff were not available (N=53), or other logistical reasons (N=33).Of the 910 patients enrolled, 212 were randomized and included in the final analysis.
Period: Overall Study
Arm/Group | Room Air | Oxygen
Started | 106 | 106
Completed | 102 | 104
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Room Air | Oxygen | Total
Number analyzed (Participants) | 102 | 104 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (5.5) | 27.2 (5.8) | 27.1 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 104 | 206
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 48 | 48 | 96
  White | 45 | 48 | 93
  Asian | 3 | 4 | 7
  Other | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 102 | 104 | 206
Insurance [Count of Participants; unit: Participants]
  Private | 48 | 46 | 94
  Public | 46 | 47 | 93
  Uninsured | 8 | 10 | 18
  Other | 0 | 1 | 1
Pre-pregnancy obesity [Count of Participants; unit: Participants] | 31 | 43 | 74
Nulliparous [Count of Participants; unit: Participants] | 56 | 59 | 115
Gestational diabetes [Count of Participants; unit: Participants] | 6 | 8 | 14
Chronic Hypertension [Count of Participants; unit: Participants] | 3 | 7 | 10
Induction of labor [Count of Participants; unit: Participants] | 71 | 78 | 149
Oxytocin [Count of Participants; unit: Participants] | 96 | 94 | 190
Epidural [Count of Participants; unit: Participants] | 97 | 99 | 196

OUTCOME MEASURES:

1. Primary Outcome: Umbilical Artery Malondialdehyde
Time Frame: At delivery
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | Room Air | Oxygen
Number analyzed (Participants) | 79 | 74
umol/L | 9.8 [6.2 to 17.4] | 10.2 [6.6 to 15.8]

2. Primary Outcome: Umbilical Artery 4-hydroxynonenal
Time Frame: At delivery
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Room Air | Oxygen
Number analyzed (Participants) | 79 | 74
pg/ml | 34.1 [10.6 to 155.2] | 29.5 [10.6 to 145]

3. Primary Outcome: Maternal Malondialdehyde
Time Frame: Within 1 hour of delivery
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Room Air | Oxygen
Number analyzed (Participants) | 80 | 79
mmol/L | 2.8 [2.1 to 3.9] | 2.5 [1.8 to 3.6]

4. Primary Outcome: Maternal 4-hydroxynonenal
Time Frame: Within 1 hour of delivery
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Room Air | Oxygen
Number analyzed (Participants) | 76 | 74
pg/ml | 190.4 [82.3 to 292.2] | 168.1 [65.9 to 312.5]

ADVERSE EVENTS:
Time Frame: 72 hours post delivery
Arm/Group | Room Air | Oxygen
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/104
Other Adverse Events (participants affected / at risk) | 5/102 | 3/104
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Room Air (N=102) | Oxygen (N=104)
Neonatal ICU stay > 72 hours (Pregnancy, puerperium and perinatal conditions) | 4 | 3
Neonatal hypothermia treatment (Pregnancy, puerperium and perinatal conditions) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/14/NCT03581214/Prot_SAP_000.pdf